CLINICAL TRIAL: NCT00345865
Title: Autologous Peripheral Blood Stem Cell Transplant for Patients With Lymphoma
Brief Title: Autologous Peripheral Stem Cell Transplant in Treating Patients With Non-Hodgkin's Lymphoma or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS048; UMN-0508M72589 (Other: IRB, University of Minnesota); UMN-MT2004-24 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma
Keywords: Hodgkin lymphoma; non-Hodgkin lymphoma; HIV-associated lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Primary Effusion | interventions — Carmustine; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor; Filgrastim; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- NHL with irradiation (Experimental): Non Hodgkin's Lymphoma patients treated with cyclophosphamide, total body irradiation therapy, peripheral blood stem cell transplantation and G-CSF.
  Interventions: Drug: cyclophosphamide; Procedure: peripheral blood stem cell transplantation; Radiation: irradiation therapy; Biological: G-CSF
- HL without irradiation (Experimental): Patients with Hodgkin's lymphoma treated with cyclosphosphamide, carmustine, etoposide, peripheral blood stem cell transplantation and G-CSF.
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Procedure: peripheral blood stem cell transplantation; Biological: G-CSF
- NHL - HIV infected with irradiation (Experimental): Non Hodgkin's Lymphoma patients infected with HIV, treated with cyclophosphamide, total body irradiation therapy, peripheral blood stem cell transplantation and G-CSF.
  Interventions: Drug: cyclophosphamide; Procedure: peripheral blood stem cell transplantation; Radiation: irradiation therapy; Biological: G-CSF
- NHL - HIV infected without irradiation (Experimental): Patients with Hodgkin's lymphoma treated with cyclosphosphamide, carmustine, etoposide, peripheral blood stem cell transplantation and G-CSF.
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Procedure: peripheral blood stem cell transplantation; Biological: G-CSF
- NHL without radiation and cyclosporine (Experimental): Patients with non Hodgkin's lymphoma ineligible to receive total body irradiation because of prior radiation and are not candidates for high dose cyclophosphamide will be treated with carmustine, etoposide, cytarabine, and melphalan followed by peripheral blood stem cell transplantation and G-CSF (called BEAM conditioning).
  Interventions: Drug: carmustine; Drug: etoposide; Procedure: peripheral blood stem cell transplantation; Biological: G-CSF; Drug: Cytarabine

INTERVENTIONS:
Drug: carmustine — Day -6, 300 mg/m^2 over 2 hour
  Other Names: BNCU
  Arms: HL without irradiation; NHL - HIV infected without irradiation; NHL without radiation and cyclosporine
Drug: cyclophosphamide — NHL with radiation: Cyclophosphamide 60 mg/kg intravenous (IV) over two hours daily x 2 days.
  HL without radiation: Cyclophosphamide, Days - 6 through -3, 1.5 gm/m^2 over 2 hours daily x 4 days.
  Cyclophosphamide will be dosed based on actual body weight (ABW) unless the patient is 20% or more of ideal body weight (IBW). If more than 20% of ideal body weight, an adjusted ideal body weight (AIBW) will be used for dosing.
  Other Names: Cytoxan
  Arms: HL without irradiation; NHL - HIV infected with irradiation; NHL - HIV infected without irradiation; NHL with irradiation
Drug: etoposide — NHL without radiation and cyclophosphamide: Etoposide 100 mg/m2 IV over 2 hours twice daily on Day -5 through -2.
  HL without radiation: 150 mg/m^2 intravenously over 4 hours every 12 hours for 6 total doses on Days -6 through -4.
  Other Names: VP-16
  Arms: HL without irradiation; NHL - HIV infected without irradiation; NHL without radiation and cyclosporine
Procedure: peripheral blood stem cell transplantation — Day 0 infuse PBSC. All patients will have PBSC collected by leukapheresis. Mobilization will be done with G-CSF alone (filgrastim) or using ifosfamide/carboplatin/etoposide and with or without rituximab. Leukapheresis is to begin on Day 5.
  Other Names: PBSC
Radiation: irradiation therapy — Patients undergo total body irradiation (TBI) twice daily on days -4 to -1.
  * > 1000 cGy to whole lung, kidney, or abdominal bath.
  * > 3000 cGy to spinal cord, myocardium, mediastinum, lumbar periaortic lymph nodes.
  * > 3600 cGy to whole brain.
  Arms: NHL - HIV infected with irradiation; NHL with irradiation
Biological: G-CSF — Day 5: Begin G-CSF 5μg/kg/day subcutaneously (SQ) rounded to the nearest vial size.
  Continue G-CSF until absolute neutrophil count (ANC) > 1500/μl x 3 consecutive days.
  If ANC falls <1000/μL, restart G-CSF.
  Other Names: filgrastim
Drug: Cytarabine — 100 mg/m^2 over one hour BID on days -6 through -2 of BEAM conditioning regimen.
  Other Names: Ara-C; cytosine arabinoside; Cytosar-U; Depocyt
  Arms: NHL without radiation and cyclosporine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide, etoposide, and carboplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored for peripheral stem cell transplant. Giving more chemotherapy, such as cyclophosphamide, carmustine, and etoposide, and total-body irradiation prepares the patient's bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy. More radiation therapy is given after transplant to kill any remaining cancer cells.

PURPOSE: This phase II trial is studying how well autologous peripheral stem cell transplant works in treating patients with non-Hodgkin's lymphoma or Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the disease-free survival and overall survival of patients with non-Hodgkin's or Hodgkin's lymphoma treated with autologous peripheral blood stem cell transplantation (PBSCT).
* Verify the safety and efficacy of autologous PBSCT in patients with HIV disease and relapsed lymphoma.

Secondary

* Evaluate immune reconstitution in HIV-positive patients undergoing autologous PBSCT and compare to immune reconstitution in HIV-negative patients.
* Predict the adequacy of peripheral blood stem cell (PBSC) harvest prior to flow analysis of a PBSC yield.
* Determine the time to engraftment for neutrophils and platelets.

OUTLINE:

* Peripheral blood stem cell (PBSC) mobilization with filgrastim (G-CSF) alone: Patients not requiring further disease reduction receive G-CSF subcutaneously (SC) once daily on days 1-8. Patients undergo PBSC collection by leukapheresis on days 5-8. Patients who do not adequately mobilize with G-CSF alone proceed to chemo-mobilization.
* Chemo-mobilization: Patients requiring further disease reduction receive 1 of 2 chemo-mobilization regimens.

  * Patients with CD20+ non-Hodgkin's lymphoma (NHL) or lymphocyte predominant Hodgkin's lymphoma: Patients receive rituximab intravenously (IV) over 6-8 hours on day 1, ifosfamide IV over 2 hours and etoposide IV over 30 minutes on days 2-4, and carboplatin IV over 1 hour on day 2. Patients receive G-CSF SC once daily beginning on day 5 and continuing until leukapheresis is completed. Patients undergo PBSC collection by leukapheresis on days 12-15.
  * All other patients: Patients receive ifosfamide IV over 2 hours and etoposide IV over 30 minutes on days 1-3 and carboplatin IV over 1 hour on day 1. Patients receive G-CSF SC once daily beginning on day 4 and continuing until leukapheresis is completed. Patients undergo PBSC collection by leukapheresis on days 12-15.
* Autologous PBSC transplantation (PBSCT) (Patients with NHL undergoing irradiation): Patients receive cyclophosphamide IV over 2 hours on days -7 and -6. Patients undergo total body irradiation (TBI) twice daily on days -4 to -1. Patients undergo autologous PBSCT on day 0. Patients receive G-CSF SC once daily beginning on day 5 and continuing until blood counts recover.
* Autologous PBSCT (Patients with Hodgkin's lymphoma or NHL not undergoing irradiation and cyclophosphamide): Patients receive camustine IV over 2 hours on days -6, etoposide IV over 2 hours twice daily on days -5 to -2, and melphalan over 1 hour on day -1. Patients undergo autologous PBSCT on day 0. Patients receive G-CSF SC once daily beginning on day 5 and continuing until blood counts recover.
* Autologous PBSC transplantation (PBSCT) (Patients with HL not undergoing irradiation): Patients receive cyclophosphamide IV over 2 hours on days -6 to -3, camustine IV over 2 hours on day -6, and etoposide IV over 4 hours twice daily on days -6 to -4. Patients undergo autologous PBSCT on day 0. Patients receive G-CSF SC once daily beginning on day 5 and continuing until blood counts recover.
* Post-transplant irradiation: Patients undergo post-transplant irradiation beginning on day 28. Persisting nodal masses ≥ 2 cm are treated with additional localized external beam irradiation.
* Post-transplant Rituximab therapy: patients with CD20+ NHL may undergo Rituximab maintenance starting between day +45 and +90 and being repeated at day +180 ± 14 days.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status: >80% (>60% if poor performance status is related to lymphoma)
* No evidence of serious organ dysfunction that is not attributable to tumor

  * Central nervous system: Patients with a history of CNS involvement by lymphoma or with relapsed primary lymphoma will be eligible.
  * Infection: Patients with serious uncontrolled infections at the time of transplant will be excluded.
* Hepatitis B: Patients who are carriers of Hepatitis B will be included in this study. These patients are not eligible to receive rituximab as a component of their chemotherapy mobilization.
* HIV disease. Patients with HIV disease are eligible for this study provided that:

  * Patients will be seen in the infectious disease (ID)/HIV clinic prior to enrollment on study for the purpose of determining eligibility and for local coordination of HIV care during the peri-transplant period.
  * Must be on a maximally active anti-HIV regimen
  * CD4+ ≥ 50/μL
  * HIV RNA viral load ≤ 100,000 copies per mL on each of samples 4 weeks apart. The most recent level must be within one month of enrollment.
* Non-Hodgkin's lymphoma (NHL). Patients with chemo-sensitive histologically confirmed NHL.

  * Precursor B-cell or Precursor T-cell NHL

    * Lymphoblastic lymphoma

      * All patients will be eligible in second or greater complete remission (CR) or first or subsequent partial remission (PR)
  * Mature B-cell Lymphomas:

    * Small lymphocytic lymphoma (SLL) or Chronic Lymphocytic Leukemia (CLL)
    * Follicular Lymphoma
    * Diffuse Large B-cell Lymphoma
    * Mantle Cell Lymphoma
    * Burkitt's/Burkitt's like
  * Mature T-cell lymphoma
* Hodgkin's lymphoma (HL)

  * patients with histologically proven HL will be eligible for transplantation after failing prior therapy.

Exclusion Criteria:

* Patients eligible for any higher priority transplant protocols
* Women who are pregnant or breast feeding
* Patients with chemotherapy resistant disease

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2005-08-24 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NHL Without Radiation and Cyclophosphamide: Patients with non Hodgkin's lymphoma ineligible to receive total body irradiation because of prior radiation and are not candidates for high dose cyclophosphamide will be treated with carmustine, etoposide, cytarabine, and melphalan followed by peripheral blood stem cell transplantation and G-CSF (called BEAM conditioning).
Period: Overall Study
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Started | 171 | 149 | 2 | 5 | 146
Completed | 171 | 149 | 2 | 5 | 146
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide | Total
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 146 | 473
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 13 | 0 | 0 | 0 | 17
  Between 18 and 65 years | 126 | 129 | 2 | 4 | 107 | 368
  >=65 years | 41 | 7 | 0 | 1 | 39 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 74 | 1 | 1 | 54 | 183
  Male | 118 | 75 | 1 | 4 | 92 | 290
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 4 | 2 | 0 | 0 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 1 | 0 | 4 | 20
  White | 147 | 127 | 1 | 5 | 135 | 415
  More than one race | 1 | 3 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 9 | 12 | 0 | 0 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 Year Progression Free Survival
Description: Progression is defined using the Response Criteria for Non-Hodgkin's Lymphoma given by NCI Sponsored International Working Group.The definition is as follows:
  At least a 50% increase from nadir of any previously identified abnormal node. Appearance of any new lesion during or at the end of therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 146
Participants | 112 | 102 | 1 | 2 | 116

2. Primary Outcome: Number of Participants With 2 Years Progression Free Survival
Description: Progression is determined using Response Criteria for Non-Hodgkin's Lymphoma given by NCI Sponsored International Working Group.
  Definition is as follows:
  At least a 50% increase from nadir of any previously identified abnormal node. Appearance of any new lesion during or at the end of therapy.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 146
Participants | 96 | 91 | 1 | 1 | 106

3. Primary Outcome: Number of Participants With 1 Year Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 146
Participants | 139 | 144 | 1 | 5 | 128

4. Primary Outcome: Number of Participants With 2 Years Overall Survival
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 146
Participants | 124 | 140 | 1 | 4 | 121

5. Secondary Outcome: Number of Participants With Hematopoietic Recovery After Transplantation
Description: return to ANC (absolute neutrophil count) more than 500 cells/milliliter.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
Number analyzed (Participants) | 171 | 149 | 2 | 5 | 145
Participants | 171 | 147 | 2 | 5 | 145

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | NHL With Irradiation | HL Without Irradiation | NHL - HIV Infected With Irradiation | NHL - HIV Infected Without Irradiation | NHL Without Radiation and Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 47/171 | 9/149 | 1/2 | 1/5 | 25/146
Serious Adverse Events (participants affected / at risk) | 34/171 | 18/149 | 1/2 | 1/5 | 0/146
Other Adverse Events (participants affected / at risk) | 125/171 | 98/149 | 2/2 | 2/5 | 120/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NHL With Irradiation (N=171) | HL Without Irradiation (N=149) | NHL - HIV Infected With Irradiation (N=2) | NHL - HIV Infected Without Irradiation (N=5) | NHL Without Radiation and Cyclophosphamide (N=146)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (12) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 12 (12) | 0 (0) | 1 (1) | 0 (0)
Pulmonary failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death due to progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death due to relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death due to multi organ failure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NHL With Irradiation (N=171) | HL Without Irradiation (N=149) | NHL - HIV Infected With Irradiation (N=2) | NHL - HIV Infected Without Irradiation (N=5) | NHL Without Radiation and Cyclophosphamide (N=146)
Infection (Infections and infestations) | 94 (331) | 63 (187) | 1 (1) | 2 (15) | 103 (291)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 67 (160) | 53 (102) | 1 (1) | 2 (6) | 55 (102)
Decreased heart function (Cardiac disorders) | 20 (26) | 16 (21) | 0 (0) | 2 (3) | 20 (31)
Neuropathy (Nervous system disorders) | 29 (39) | 12 (13) | 0 (0) | 0 (0) | 14 (16)
Other Kidney disorder (Renal and urinary disorders) | 23 (36) | 6 (10) | 1 (2) | 2 (2) | 9 (10)
sensory loss (Nervous system disorders) | 20 (26) | 4 (4) | 0 (0) | 0 (0) | 8 (8)
Deep vein thrombosis (Vascular disorders) | 9 (10) | 8 (9) | 1 (1) | 0 (0) | 15 (16)
Intubation (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 6 (8) | 0 (0) | 0 (0) | 6 (7)
Thrombosis (Vascular disorders) | 10 (10) | 8 (9) | 1 (1) | 0 (0) | 8 (10)
GI bleeding (Gastrointestinal disorders) | 12 (13) | 3 (4) | 1 (1) | 1 (2) | 5 (6)
deconditioning (Metabolism and nutrition disorders) | 7 (11) | 2 (2) | 0 (0) | 0 (0) | 7 (9)
Surgery (Injury, poisoning and procedural complications) | 5 (8) | 3 (3) | 0 (0) | 1 (1) | 5 (6)
hypothyroidism (Endocrine disorders) | 9 (10) | 10 (11) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT00345865/Prot_SAP_000.pdf